CLINICAL TRIAL: NCT06676995
Title: Parkinson's Disease: Overall Symptoms Improvement With Transcranial Pulse Stimulation (TPS)
Brief Title: Effects of Transcranial Pulse Stimulation in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Felipe Fregni, MD, PhD, MPH, Director of the Neuromodulation Center, Professor of Rehabilitation, Spaulding Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024P002627
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Parkinson
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- TPS (Experimental)
  Interventions: Device: Transcranial Pulse Stimulation (TPS)

INTERVENTIONS:
Device: Transcranial Pulse Stimulation (TPS) — Transcranial Pulse Stimulation (TPS) is a non invasive brain stimulation technology that applies repetitive single high-pressure ultrashort shockwave pulses within the ultrasound frequency range to stimulate the brain. Subjects will receive 12 TPS sessions conducted three times weekly, for about 40 to 50 minutes/day, over four consecutive weeks.

SUMMARY:
The investigators are studying if Transcranial Pulse Stimulation (TPS) can improve various symptoms, including movement problems, thinking abilities, mood, fatigue, freezing while walking, voice quality, and issues with smell and taste. Previous research suggests TPS might help in Alzheimer's disease and could be helpful for Parkinson's as well. Investigators will check if TPS is safe, practical, and if it makes a noticeable difference in these symptoms compared to before the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of "probable" or "possible" PD, as defined by the current clinical criteria (52) or as confirmed by a co-investigator neurologist or confirmation via medical records or a letter from a patient's physician.
2. Age from 40 to 90 years old.
3. Disease stages 2 to 4 based on the UPDRS scale subdomain V (or Hoehn and Yahr scale).
4. Taking stable medications for PD for at least 30 days.

Exclusion Criteria:

1. Features suggestive of other causes of parkinsonism/Parkinson's-plus syndromes.
2. History of deep brain stimulation, brain ablation surgeries, or malignant mass brain lesions.
3. History of schizophrenia, bipolar illness, or alcohol/drug abuse within the past six months.
4. Need for rapid clinical response due to conditions such as initiation, psychosis, or suicidality.
5. Contraindications to transcranial brain stimulation (i.e., metal objects in the head, metal implanted brain medical devices, cortisone treatments within six weeks before the first stimulation session, CNS thrombosis, etc).
6. Unstable medical conditions (e.g., uncontrolled diabetes, uncompensated cardiac issues, heart failure, uncompensated pulmonary disease, or chronic obstructive pulmonary disease).
7. Contraindications to MRI according to MGB screening in the Martinos-Center (i.e., pacemaker, defibrillator or wires other than sternal wires, metallic foreign body in the eye, or drug infusion devices - if the models of these devices are not compatible with MRI).
8. Pregnancy.
9. Epilepsy or disorders that significantly increase the likelihood of seizures, including: (i) severe traumatic brain injury; (ii) congenital birth defects leading to seizures; (iii) brain tumor; (iv) metabolic disorders associated with seizures; (v) intracranial or subarachnoid hemorrhage; and (vi) non-lacunar strokes.
10. Bed- or wheelchair-bound patients.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-12-31 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS) | Baseline, post intervention (from enrollment to the end of intervention at 4 weeks), and follow up (after 4 weeks from the last day of intervention).)
  Unified Parkinson's Disease Rating Scale (UPDRS) evaluates the motor function, non-motor symptoms (mentation, behavior, and mood), activities of daily living, and complications of therapy. Each item has 0-4 ratings: 0 (normal), 1 (slight), 2 (mild), 3 (moderate), and 4 (severe). The total score can be up to 232.

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Rehabilitation Hospital, Cambridge, Massachusetts, United States

REFERENCES:
- [Background] Shinzato GT, Assone T, Sandler PC, Pacheco-Barrios K, Fregni F, Radanovic M, Forlenza OV, Battistella LR. Non-invasive sound wave brain stimulation with Transcranial Pulse Stimulation (TPS) improves neuropsychiatric symptoms in Alzheimer's disease. Brain Stimul. 2024 Mar-Apr;17(2):413-415. doi: 10.1016/j.brs.2024.03.007. Epub 2024 Mar 20. PMID 38513821
- [Background] Fong TKH, Cheung T, Ngan STJ, Tong K, Lui WYV, Chan WC, Wong CSM, Cheng CPW. Transcranial pulse stimulation in the treatment of mild neurocognitive disorders. Ann Clin Transl Neurol. 2023 Oct;10(10):1885-1890. doi: 10.1002/acn3.51882. Epub 2023 Aug 21. PMID 37607114
- [Background] Osou S, Radjenovic S, Bender L, Gaal M, Zettl A, Dorl G, Matt E, Beisteiner R. Novel ultrasound neuromodulation therapy with transcranial pulse stimulation (TPS) in Parkinson's disease: a first retrospective analysis. J Neurol. 2024 Mar;271(3):1462-1468. doi: 10.1007/s00415-023-12114-1. Epub 2023 Nov 30. PMID 38032371